CLINICAL TRIAL: NCT01078532
Title: Self Management & Reminders With Technology: SMART Appraisal of an Integrated Personal Health Record (SMART PHR)
Brief Title: Self Management and Reminders With Technology: SMART Appraisal of an Integrated Personal Health Record (PHR)
Acronym: SMART PHR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HS018167
Record Dates: First submitted 2010-02-27; First posted 2010-03-02 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Cardiovascular Risk
Keywords: medically complex diseases that increase cardiovascular risk

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMART PHR (Experimental): Patients receive the active PHR
  Interventions: Other: SMART PHR
- Passive PHR (Other): Usual PHR Care
  Interventions: Other: usual care

INTERVENTIONS:
Other: SMART PHR — Patient receives an active PHR
  Arms: SMART PHR
Other: usual care — Usual passive PHR
  Arms: Passive PHR

SUMMARY:
This project seeks to improve health care outcomes in complex patients with cardiovascular disease (CVD) or who are at high risk for developing CVD by promoting patient self-management. This will be accomplished in 4 diverse, large primary care practices through the following 3 aims: (1) develop a patient-specific, active component to an existing electronic PHR directed towards patients with complex illnesses that is designed to reduce the risk of cardiovascular disease, (2) conduct a randomized controlled trial of the effectiveness of passive and active PHRs for improving adherence and clinical outcomes of complex patients in an ambulatory environment, and (3) enumerate the barriers and facilitators to implementation and use of an PHR among providers and patients in an ambulatory setting. To accomplish the aim 1, a users group will be assembled to determine which potential features of an 'active PHR' would be most acceptable and useful to them. To accomplish the 2nd aim, 1,000 patients with complex chronic disease leading to increased cardiovascular risk (i.e., CVD or 2 of the 4 conditions of hypertension (HTN), diabetes mellitus (DM), or hyperlipidemia requiring at least one medication for control) will be randomized to a passive PHR (n=500), or an active PHR (n=500) at 4 sites where the PHR currently is installed and in use. Outcomes to be assessed include improvement in control of risk factors (e.g., blood pressure), frequency of compliance with testing guidelines (e.g., annual dilated retinal exams in DM), and clinical outcomes (e.g., myocardial infarction, hospitalizations). Aim 3 will be accomplished by surveying all participants using the PHR, along with nurses and physicians at the study sites, and by conducting focus groups of PHR participants, nurses, and physicians to determine the most useful features of the PHR and to barriers and facilitators of use.

ELIGIBILITY:
Inclusion Criteria:

* >=18, if they have medically complex diseases that increase cardiovascular risk not yet a PHR user

Exclusion Criteria:

* current PHR user life-expectancy of less than 6 months dementia or disability that prevents them from being able to utilize a PHR (such as blindness)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1815 (Actual)
Dates: Start 2010-04; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
improved targeted chronic disease outcomes | 1 year
  blood pressure and low density lipoprotein level (LDL) in all patients, and A1C in patients who have diabetes. For patients on medications requiring monitoring of electrolytes and creatinine, we will look at changes in these parameters as well.

SECONDARY OUTCOMES:
change in value in these outcome measures (lipid levels, blood pressure, and A1c levels) | 1 year
rates of adherence to diagnostic and therapeutic recommendations | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Roberts, MD, MPP, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Primary Care practices, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Hess R, Fischer GS, Sullivan SM, Dong X, Weimer M, Zeith C, Clark S, Roberts MS. Patterns of response to patient-centered decision support through a personal health record. Telemed J E Health. 2014 Nov;20(11):984-9. doi: 10.1089/tmj.2013.0332. Epub 2014 Sep 22. PMID 25243350